CLINICAL TRIAL: NCT00920114
Title: Estimate of the Activity and the Forecast of the Lupus Disease of the Adult by a Transcriptomic Score (STUDY LU-PUCE)
Acronym: LU-PUCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Assistance Publique Hopitaux De Marseille, Direction de la recherche
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2009/04; 2009-A00257-50
Record Dates: First submitted 2009-06-05; First posted 2009-06-15 (Estimated); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Lupus Disease
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Lupus disease (Experimental)
  Interventions: Biological: blood sample
- Healthy witnesses (Active Comparator)
  Interventions: Biological: blood sample
- Healthy witnesses with an other auto-immune disease (Active Comparator)
  Interventions: Biological: blood sample

INTERVENTIONS:
Biological: blood sample

SUMMARY:
Lupus erythematosus systemic is an auto-immune disease the evaluation of the activity of which remains very difficult because of an heterogeneousness of the clinical and biological symptoms. The aim of this study is to develop objective, specific and not invasive methods of evaluation of the activity and the forecast of the disease by using an analysis of the transcriptome on circulating blood. A transcriptomic analysis will be realized in parallel by the usual clinico-biological follow-up at the patients affected by systemic lupus, while the diagnosis before treatment, then during every revaluation of the disease during the period of the study. The already treated patients can also be included in this study.

ELIGIBILITY:
Inclusion Criteria:

* Lupus disease diagnosed for lupus disease arm
* Signed assent

Exclusion Criteria:

* non-compliance
* pregnancy
* persons without social coverage

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2009-05; Primary Completion 2011-05 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Identify the genes expressed during the disease to allow the calculation of a transcriptomic score and study the correlation of this transcriptionnal score with the SLEDAI score | 2 years

SECONDARY OUTCOMES:
Identify genes correlated in various histological classes of lupus renal disease and types of pushes of the disease; to allow the calculation of a transcriptomic score and its correlation with the BILAG score | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Laurent CHICHE, Principal Investigator — Assistance Publique-Hôpitaux de Marseille
Locations (1):
- Assistance Publique-Hopitaux de Marseille, Marseille, France

REFERENCES:
- [Background] Jourde-Chiche N, Whalen E, Gondouin B, Speake C, Gersuk V, Dussol B, Burtey S, Pascual V, Chaussabel D, Chiche L. Modular transcriptional repertoire analyses identify a blood neutrophil signature as a candidate biomarker for lupus nephritis. Rheumatology (Oxford). 2017 Mar 1;56(3):477-487. doi: 10.1093/rheumatology/kew439. PMID 28031441
- [Background] Bettacchioli E, Chiche L, Chaussabel D, Cornec D, Jourde-Chiche N, Rinchai D. An interactive web application for exploring systemic lupus erythematosus blood transcriptomic diversity. Database (Oxford). 2024 May 28;2024:baae045. doi: 10.1093/database/baae045. PMID 38805754
- [Background] Arcani R, Jouve E, Chiche L, Jourde-Chiche N. Categorization of patients with systemic lupus erythematosus using disease activity, patient-reported outcomes, and transcriptomic signatures. Clin Rheumatol. 2023 Jun;42(6):1555-1563. doi: 10.1007/s10067-023-06525-8. Epub 2023 Feb 10. PMID 36759402
- [Background] Seguier J, Jouve E, Bobot M, Whalen E, Dussol B, Gentile S, Burtey S, Halfon P, Retornaz F, Chaussabel D, Chiche L, Jourde-Chiche N. Paradoxical association between blood modular interferon signatures and quality of life in patients with systemic lupus erythematosus. Rheumatology (Oxford). 2020 Aug 1;59(8):1975-1983. doi: 10.1093/rheumatology/kez541. PMID 31776548
- [Result] Chiche L, Jourde-Chiche N, Whalen E, Presnell S, Gersuk V, Dang K, Anguiano E, Quinn C, Burtey S, Berland Y, Kaplanski G, Harle JR, Pascual V, Chaussabel D. Modular transcriptional repertoire analyses of adults with systemic lupus erythematosus reveal distinct type I and type II interferon signatures. Arthritis Rheumatol. 2014 Jun;66(6):1583-95. doi: 10.1002/art.38628. PMID 24644022